CLINICAL TRIAL: NCT02800252
Title: Effects of Omega-3 Polyunsaturated Fatty Acids Daily Supplementation Plus Low-dose Aspirin as Adjunct to Full-mouth Periodontal Ultrasonic Debridement for the Treatment of Chronic Periodontitis in Type 2 Diabetics: Randomized Clinical Trial
Brief Title: Effects of Omega-3 Plus Low-dose Aspirin as Adjunct to Periodontal Debridement for Chronic Periodontitis in Diabetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Nídia Cristina Castro dos Santos, DDS, MS, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCSFOSJC
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus; Chronic Periodontitis
Keywords: fatty acids; aspirin; diabetes mellitus; chronic periodontitis; periodontal debridement
MeSH Terms: conditions — Diabetes Mellitus; Chronic Periodontitis | interventions — Docosahexaenoic Acids; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Placebo Comparator): Full-mouth periodontal debridement and placebo
  Interventions: Drug: Placebo
- Test 1 (Active Comparator): Full-mouth periodontal debridement, 3g omega-3 plus 100mg aspirin daily for 60 days after periodontal therapy
  Interventions: Drug: 3g omega-3 plus 100mg aspirin daily for 60 days
- Test 2 (Active Comparator): omega-3 plus aspirin before periodontal therapy
  Interventions: Drug: omega-3 plus aspirin before periodontal therapy

INTERVENTIONS:
Drug: Placebo — One-stage full-mouth periodontal ultrasonic debridement plus placebo intervention
  Arms: Control Group
Drug: 3g omega-3 plus 100mg aspirin daily for 60 days — Full-mouth periodontal debridement, 3g omega-3 plus 100mg aspirin daily for 60 days after periodontal therapy
  Other Names: omega-3 polyunsaturated fatty acids; acetylsalicylic acid
  Arms: Test 1
Drug: omega-3 plus aspirin before periodontal therapy — Full-mouth periodontal debridement, 3g omega-3 plus 100mg aspirin daily for 60 days before periodontal therapy
  Other Names: omega-3 polyunsaturated fatty acids; acetylsalicylic acid
  Arms: Test 2

SUMMARY:
Therefore, the aim of this study is to investigate the effectiveness of daily supplementation of omega-3 polyunsaturated fatty acids and low-dose aspirin as adjunct therapy to one-stage full-mouth periodontal ultrasonic debridement for the treatment of chronic periodontitis in type 2 diabetic patients through a superiority randomized clinical trial.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) has become a global epidemic. Its complications can have a significant impact on quality of life, longevity, and costs in public health. The World Health Organization (WHO) estimates that by 2040, 642 million people will suffer from diabetes, around 10% of the world adult population (WHO, 2015). Periodontal Diseases are considered the sixth complication of DM. This close relationship between both diseases is characterized by mutual influence. Thus, an appropriate control of periodontal disease may facilitate the DM control, improving quality of life on diabetic patients. Besides that, the presence of DM might impair prognosis of diverse dental treatments due to its inflammatory nature, negative influence on wound healing, on bone biology, and the establishment of infections. As a host modulatory therapy (HMT), the daily supplementation of omega-3 polyunsaturated fatty acids and low-dose aspirin has been proposed as adjunct therapy to the treatment of chronic periodontitis, showing good clinical and metabolic results in normoglycemic patients. Therefore, the aim of this study is to investigate the effectiveness of daily supplementation of omega-3 polyunsaturated fatty acids and low-dose aspirin as adjunct therapy to one-stage full-mouth periodontal ultrasonic debridement for the treatment of chronic periodontitis in type 2 diabetic patients through a superiority randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* a) Age ≥35 b) diagnosis of type 2 DM for ≥5 years c) DM treatment with oral hypoglycemic agents or insulin supplementation and diet d) glycated hemoglobin (HbA1c) levels from 6.5% to 11% e) at least 15 teeth (excluding third molars and teeth indicated for extraction) f) moderate to severe generalized chronic periodontitis (Armitage, 1999) g) agree and sign the formal consent to participate in the study after receiving an explanation of risks and benefits from an individual who is not a member of the study (Resolution number 196 - October, 1996, and Ethics and Code of Professional Conduct in Dentistry - CFO179/93).

Exclusion Criteria:

* a) medical conditions that required prophylactic antimicrobial coverage b) scaling and root planing in the previous 6 months c) antimicrobial therapies in the previous 6 months d) anti-inflammatory therapies in the previous 6 months e) systemic conditions, other than DM, that could affect the progression of chronic periodontitis f) current use of medication that could interfere with periodontal response to treatment g) pregnancy or lactation h) smoking

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Periodontal pockets with mean probing depth (PD) ≥5mm | Baseline, 90 days, 180 days

SECONDARY OUTCOMES:
Probing depth (mm) | Baseline, 90 days, 180 days
  Using a manual periodontal probe (North Carolina, HuFriedy, Chicago, IL, USA)
Clinical attachment level (mm) | Baseline, 90 days, 180 days
  Using a manual periodontal probe (North Carolina, HuFriedy, Chicago, IL, USA)
Gingival recession (mm) | Baseline, 90 days, 180 days
  Using a manual periodontal probe (North Carolina, HuFriedy, Chicago, IL, USA)
Bleeding on probing (%) | Baseline, 90 days, 180 days
  Using a manual periodontal probe (North Carolina, HuFriedy, Chicago, IL, USA)
Plaque index (%) | Baseline, 90 days, 180 days
  Using a manual periodontal probe (North Carolina, HuFriedy, Chicago, IL, USA)

OTHER OUTCOMES:
Glycated hemoglobin | Baseline, 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Study Director — UPECLIN HC FM Botucatu Unesp
Locations (1):
- UNESP, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] El-Sharkawy H, Aboelsaad N, Eliwa M, Darweesh M, Alshahat M, Kantarci A, Hasturk H, Van Dyke TE. Adjunctive treatment of chronic periodontitis with daily dietary supplementation with omega-3 Fatty acids and low-dose aspirin. J Periodontol. 2010 Nov;81(11):1635-43. doi: 10.1902/jop.2010.090628. Epub 2010 Jun 23. PMID 20572767
- [Derived] Castro Dos Santos N, Mangussi A, Ribeiro T, Silva RNB, Santamaria MP, Feres M, VAN Dyke T, Lorena AC. Factors influencing the response to periodontal therapy in patients with diabetes: post hoc analysis of a randomized clinical trial using machine learning. J Appl Oral Sci. 2025 Jul 25;33:e20250211. doi: 10.1590/1678-7757-2025-0211. eCollection 2025. PMID 40736087
- [Derived] Dos Santos NC, Araujo CF, Andere NMRB, Miguel MMV, Westphal MRA, Van Dyke T, Santamaria MP. Omega-3 Fatty Acids and Low-Dose Aspirin in the Treatment of Periodontitis and Metabolic Syndrome: Case Report. J Int Acad Periodontol. 2020 Oct 1;22(4):223-230. PMID 32980834